CLINICAL TRIAL: NCT01040364
Title: Incidence of Internal Hernias After Laparoscopic Roux-en-Y Gastric Bypass Over the Last Decade: 1997 to 2008
Brief Title: Internal Hernias After Laparoscopic Gastric Bypass
Acronym: IHafterLRYGB
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: CMC IRB No. 2009024; U1111-1113-0414 (Other: World Health Organization, Universal Trial Number)
Record Dates: First submitted 2009-12-26; First posted 2009-12-29 (Estimated); Last update posted 2013-09-24 (Estimated); Status verified 2013-09

CONDITIONS: Internal Hernia; Mesocolic Hernia; Petersen´s Hernia; Jejunojejunostomy Hernia; Bowel Obstruction; Ischemic Bowel
Keywords: Internal hernia; Mesocolic hernia; Petersen´s hernia; Jejunojejunostomy hernia; Bowel obstruction; Ischemic bowel; Complication after gastric bypass; Re-operative bariatric surgery; Chronic pain after gastric bypass
MeSH Terms: conditions — Internal Hernia; Intestinal Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Interna hernia after primary gastric bypass

SUMMARY:
The main goal of this study is to describe the trends in the incidence rate of internal hernia presentation after different modifications of the mesenteric closure technique after primary laparoscopic Roux-en-Y gastric bypass (RYGB) surgery from 1997-2009.

DETAILED DESCRIPTION:
The main goal of this study is to describe and analyze the trends in the incidence rate of internal hernia presentation after different modifications of the mesenteric closure technique after Primary Laparoscopic RYGB Surgery from 1997 to 2009.

Secondary study aims are to describe the following points 1. Clinical presentation, whether acute (small bowel obstruction), chronic (intermittent abdominal pain), or incidental finding -(asymptomatic); 2. Preoperative image studies. The percentage of patients that underwent preoperative CT/contrast studies as well as the percentage of patients that had positive, undetermined, and normal results; 3. Site of internal herniation including transverse mesocolon, jejunal mesentery, and Peterson's space as well as single vs. multiple internal hernias. This study along with the existing literature will allow us to formulate preliminary clinical recommendations.

This research is in line with the most current provocative new ideas and recent high impact publications. Most literature points towards the antecolic routing of the Roux limb to decrease the incidence rate of internal hernia formation. However, with this study we will demonstrate the statistically and clinically significant decrement of internal hernia formation with the improvement of the closure technique with a retrocolic antegastric routing of the Roux limb.

The epidemic of overweight and obesity in the United States of America along with its comorbidities continues to expand. Bariatric surgery has demonstrated to be the most effective and sustained method to control severe obesity and its comorbidities. For instance, type 2 diabetes mellitus was completely resolved in 76.8 percent, systemic arterial hypertension was resolved in 61.7 percent, dyslipidemia improved in 70 percent, and obstructive sleep apnea-hypopnea syndrome was resolved in 85.7 percent. Furthermore, bariatric surgery significantly increases life expectancy (89 percent) and decreases overall mortality (30 to 40 percent), particularly deaths from diabetes, heart disease, and cancer. Lastly, preliminary evidence about downstream savings associated with bariatric surgery offset the initial costs in 2 to 4 years.

Since 1998, there has been a substantially progressive increase in bariatric surgery. In 2005, the American Society of Metabolic and Bariatric Surgery "ASMBS" reported that 81 percent of bariatric procedures were approached laparoscopically. 205,000 people, in 2007, had bariatric surgery in the United States from which approximately 80 percentage of these were Gastric Bypass. Moreover, there is a mismatch between eligibility and receipt of bariatric surgery with just less than 1% of the eligible population being treated for morbid obesity through bariatric surgery10. Along with the increasing number of elective primary weight loss procedures, up to 20 percent of post RYGB patients cannot sustain their weight loss beyond 2 to 3 years after the primary bariatric procedure11. Thus, revisional surgery for poor weight loss and reoperations for technical or mechanical complications will rise in a parallel manner. RYGB is consistently considered the revisional procedure of choice for failed restrictive procedures.

At present there are three broad categories of bariatric procedures according to its mechanism of action 1. purely restrictive, 2. primarily restrictive with some malabsorption, and 3. primarily malabsorptive with some restriction. Modern standard bariatric procedures recognized by the American Society for Metabolic and Bariatric Surgery "ASMBS" include the following 1. adjustable gastric band, 2. sleeve gastrectomy, 3. gastric bypass, 4. biliopancreatic diversion, and 5. duodenal switch.

There are no multi center, randomized, double blinded control trials comparing the different standard bariatric procedures. Gastric bypass is the oldest available bariatric procedure; without any randomized controlled trials, it is considered the gold standard procedure in the United States.

Incisional hernias occur at a higher incidence rate after open RYGB, approximately 20 percent, whereas after laparoscopic Roux-en-Y gastric bypass "RYGB", the incidence rate is very low. Conversely, Internal hernia is a rare complication with the open approach whereas after laparoscopic RYGB the incidence rate has been reported somewhere between 0.2 to 8.6 percent. The most accepted theory is due to decreased adhesion formation after laparoscopic surgery compared to open surgery.

Other factors associated with a higher incidence of internal hernia formation after RYGB are 1. childbearing age with the consequent pregnancy after RYGB, 2. Roux limb routing, 3. Closure of mesenteric and or mesocolic defects.

Although there have been no randomized controlled trials comparing different techniques of laparoscopic RYGB, several authors have report lower rates after modifying their technique from a retrocolic to an antecolic approach. On the other hand, others support meticulous defect closure as the most important factor in reducing hernia formation.

The method of fixation and mesenteric closure has evolved. Initially, as with the open approach, defects were not closed. Then, absorbable sutures were used which were changed for interrupted non-absorbable sutures. Lastly, continuous non-absorbable material for closing all defects was recommended by Sugerman.

Summarizing, there is no high level of evidence for recommending the best strategy to decrease the incidence rate the potentially devastating complication of internal hernia after laparoscopic RYGB. After reviewing the literature the trend is toward lower rates of internal hernia formation with antecolic compared to retrocolic, and with defect closure compared to nonclosure. There is great variation in the incidence rate among the reported series reflecting incomplete follow-up and other factors may affect outcomes. With this study, we will analyze the trends in the incidence rate of internal hernia formation among different subgroups in our consecutive series of more than 7,500 laparoscopic retrocolic RYGB with a hand-sawn gastrojejunostomy. With this consecutive series, we will confirm reports of small series that meticulous closure technique of mesocolic/mesenteric defects with continuous nonabsorbable material clinically and statistically decreases the formation rate of internal hernias after laparoscopic gastric bypass.

ELIGIBILITY:
Inclusion Criteria:

* patient status post primary laparoscopic standard RYGB surgery who underwent internal hernia reduction and repair with any or the combination of the following:

  * closure of synchronous mesocolic or mesenteric space defects without incarcerated bowel
  * conversion to open (laparotomy)
  * small bowel resection with or without reversal
* status post primary laparoscopic standard RYGB surgery with incidental finding of internal hernia space defect with or without bowel through the defect

Exclusion Criteria:

* any other type of re-operative surgery after primary standard RYGB
* patient age < 18 years
* missing records and/or unreachable patients with scant information for analysis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with internal hernia after different modifications of the mesenteric closure technique after Primary Laparoscopic RYGB surgery from 1997-2009.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2009-05; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Closure technique for mesocolic defect: 1- non-closure, 2- running with absorbable material, 3- interrupted with non-absorbable material, and 4- running with non-absorbable | throughout follow-up
recurrence of symptomatic mesocolic internal hernia | throughout follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Francisco M Tercero, MD, Study Director — Research Associate, University of California San Francisco; Kelvin D Higa, MD, Principal Investigator — Professor of Surgery, University of California San Francisco
Locations (1):
- UCSF Fresno Center for Medical Education and Research, Department of Surgery, Fresno, California, United States

REFERENCES:
- [Background] Higa KD, Boone KB, Ho T, Davies OG. Laparoscopic Roux-en-Y gastric bypass for morbid obesity: technique and preliminary results of our first 400 patients. Arch Surg. 2000 Sep;135(9):1029-33; discussion 1033-4. doi: 10.1001/archsurg.135.9.1029. PMID 10982506
- [Background] McTigue KM, Harris R, Hemphill B, Lux L, Sutton S, Bunton AJ, Lohr KN. Screening and interventions for obesity in adults: summary of the evidence for the U.S. Preventive Services Task Force. Ann Intern Med. 2003 Dec 2;139(11):933-49. doi: 10.7326/0003-4819-139-11-200312020-00013. PMID 14644897
- [Background] Buchwald H, Avidor Y, Braunwald E, Jensen MD, Pories W, Fahrbach K, Schoelles K. Bariatric surgery: a systematic review and meta-analysis. JAMA. 2004 Oct 13;292(14):1724-37. doi: 10.1001/jama.292.14.1724. PMID 15479938
- [Background] Christou NV, Sampalis JS, Liberman M, Look D, Auger S, McLean AP, MacLean LD. Surgery decreases long-term mortality, morbidity, and health care use in morbidly obese patients. Ann Surg. 2004 Sep;240(3):416-23; discussion 423-4. doi: 10.1097/01.sla.0000137343.63376.19. PMID 15319713
- [Background] Adams TD, Gress RE, Smith SC, Halverson RC, Simper SC, Rosamond WD, Lamonte MJ, Stroup AM, Hunt SC. Long-term mortality after gastric bypass surgery. N Engl J Med. 2007 Aug 23;357(8):753-61. doi: 10.1056/NEJMoa066603. PMID 17715409
- [Background] Sjostrom L, Narbro K, Sjostrom CD, Karason K, Larsson B, Wedel H, Lystig T, Sullivan M, Bouchard C, Carlsson B, Bengtsson C, Dahlgren S, Gummesson A, Jacobson P, Karlsson J, Lindroos AK, Lonroth H, Naslund I, Olbers T, Stenlof K, Torgerson J, Agren G, Carlsson LM; Swedish Obese Subjects Study. Effects of bariatric surgery on mortality in Swedish obese subjects. N Engl J Med. 2007 Aug 23;357(8):741-52. doi: 10.1056/NEJMoa066254. PMID 17715408
- [Background] Cremieux PY, Buchwald H, Shikora SA, Ghosh A, Yang HE, Buessing M. A study on the economic impact of bariatric surgery. Am J Manag Care. 2008 Sep;14(9):589-96. PMID 18778174
- [Background] Santry HP, Gillen DL, Lauderdale DS. Trends in bariatric surgical procedures. JAMA. 2005 Oct 19;294(15):1909-17. doi: 10.1001/jama.294.15.1909. PMID 16234497
- [Background] Flum DR, Khan TV, Dellinger EP. Toward the rational and equitable use of bariatric surgery. JAMA. 2007 Sep 26;298(12):1442-4. doi: 10.1001/jama.298.12.1442. No abstract available. PMID 17895461
- [Background] Meguid MM, Glade MJ, Middleton FA. Weight regain after Roux-en-Y: a significant 20% complication related to PYY. Nutrition. 2008 Sep;24(9):832-42. doi: 10.1016/j.nut.2008.06.027. PMID 18725080
- [Background] Nguyen NT. Reoperations and revisions in bariatric surgery. Surg Endosc. 2007 Nov;21(11):1907-8. doi: 10.1007/s00464-007-9572-6. Epub 2007 Sep 8. No abstract available. PMID 17828427
- [Background] http://www.asbs.org/htm/Private/resolution.html. American Society of Metabolic and Bariatric Surgeons.
- [Background] Capella RF, Iannace VA, Capella JF. Bowel obstruction after open and laparoscopic gastric bypass surgery for morbid obesity. J Am Coll Surg. 2006 Sep;203(3):328-35. doi: 10.1016/j.jamcollsurg.2006.05.301. Epub 2006 Jul 27. PMID 16931305
- [Background] Champion JK, Williams M. Small bowel obstruction and internal hernias after laparoscopic Roux-en-Y gastric bypass. Obes Surg. 2003 Aug;13(4):596-600. doi: 10.1381/096089203322190808. PMID 12935361
- [Background] Felsher J, Brodsky J, Brody F. Small bowel obstruction after laparoscopic Roux-en-Y gastric bypass. Surgery. 2003 Sep;134(3):501-5. doi: 10.1067/s0039-6060(03)00251-4. PMID 14555940
- [Background] Hwang RF, Swartz DE, Felix EL. Causes of small bowel obstruction after laparoscopic gastric bypass. Surg Endosc. 2004 Nov;18(11):1631-5. doi: 10.1007/s00464-004-8804-2. Epub 2004 Oct 11. PMID 15931476
- [Background] Carmody B, DeMaria EJ, Jamal M, Johnson J, Carbonell A, Kellum J, Maher J. Internal hernia after laparoscopic Roux-en-Y gastric bypass. Surg Obes Relat Dis. 2005 Nov-Dec;1(6):543-8. doi: 10.1016/j.soard.2005.08.005. Epub 2005 Sep 28. PMID 16925288
- [Background] Cho M, Pinto D, Carrodeguas L, Lascano C, Soto F, Whipple O, Simpfendorfer C, Gonzalvo JP, Zundel N, Szomstein S, Rosenthal RJ. Frequency and management of internal hernias after laparoscopic antecolic antegastric Roux-en-Y gastric bypass without division of the small bowel mesentery or closure of mesenteric defects: review of 1400 consecutive cases. Surg Obes Relat Dis. 2006 Mar-Apr;2(2):87-91. doi: 10.1016/j.soard.2005.11.004. Epub 2006 Mar 3. PMID 16925328
- [Background] DeMaria EJ, Sugerman HJ, Kellum JM, Meador JG, Wolfe LG. Results of 281 consecutive total laparoscopic Roux-en-Y gastric bypasses to treat morbid obesity. Ann Surg. 2002 May;235(5):640-5; discussion 645-7. doi: 10.1097/00000658-200205000-00005. PMID 11981209
- [Background] Dresel A, Kuhn JA, Westmoreland MV, Talaasen LJ, McCarty TM. Establishing a laparoscopic gastric bypass program. Am J Surg. 2002 Dec;184(6):617-20; discussion 620. doi: 10.1016/s0002-9610(02)01098-x. PMID 12488190
- [Background] Eckhauser A, Torquati A, Youssef Y, Kaiser JL, Richards WO. Internal hernia: postoperative complication of roux-en-Y gastric bypass surgery. Am Surg. 2006 Jul;72(7):581-4; discussion 584-5. PMID 16875078
- [Background] Filip JE, Mattar SG, Bowers SP, Smith CD. Internal hernia formation after laparoscopic Roux-en-Y gastric bypass for morbid obesity. Am Surg. 2002 Jul;68(7):640-3. PMID 12132750
- [Background] Garza E Jr, Kuhn J, Arnold D, Nicholson W, Reddy S, McCarty T. Internal hernias after laparoscopic Roux-en-Y gastric bypass. Am J Surg. 2004 Dec;188(6):796-800. doi: 10.1016/j.amjsurg.2004.08.049. PMID 15619502
- [Background] Gould JC, Garren MJ, Boll V, Starling JR. Laparoscopic gastric bypass: risks vs. benefits up to two years following surgery in super-super obese patients. Surgery. 2006 Oct;140(4):524-9; discussion 529-31. doi: 10.1016/j.surg.2006.07.002. PMID 17011899
- [Background] Higa KD, Ho T, Boone KB. Internal hernias after laparoscopic Roux-en-Y gastric bypass: incidence, treatment and prevention. Obes Surg. 2003 Jun;13(3):350-4. doi: 10.1381/096089203765887642. PMID 12841892
- [Background] Hedley AA, Ogden CL, Johnson CL, Carroll MD, Curtin LR, Flegal KM. Prevalence of overweight and obesity among US children, adolescents, and adults, 1999-2002. JAMA. 2004 Jun 16;291(23):2847-50. doi: 10.1001/jama.291.23.2847. PMID 15199035
- See also: "Click here for more information about the department sponsor´s web site" — http://www.fresno.ucsf.edu/surgery